CLINICAL TRIAL: NCT07150780
Title: Benefits of no FASTing Prior to Elective Cardiac CATHeterization (FAST CATH): A Single-center Randomized-controlled Trial Comparing a Non-fasting Pre-procedure Approach to the Standard of Care in Adults Undergoing Elective Cardiac Catheterization With Moderate Sedation
Brief Title: Benefits of no Fasting Compared to Fasting Prior to Elective Cardiac Catheterization: A Single-center Randomized-controlled Trial
Acronym: FAST CATH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Munson Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MHCIIR001-2025
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease; Cardiac Catheterization; Cardiac Diseases
Keywords: Cardiac catheterization; Fasting; Patient Satisfaction
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases; Fasting; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting (No Intervention): Prior to the subjects elective cardiac catheterization, they will be instructed to fast for 6 hours with the allowance of clear liquids up to 2 hours.
- Non-fasting (Experimental): Subjects will be instructed to continue to eat and drink according to their normal diet without restriction, prior to their cardiac catheterization.
  Interventions: Procedure: Pre-operative instructions to eat and drink at liberty

INTERVENTIONS:
Procedure: Pre-operative instructions to eat and drink at liberty — Subjects will be instructed to eat and drink at liberty prior to their schedule elective cardiac catheterization.
  Arms: Non-fasting

SUMMARY:
More than one million cardiac catheterizations (CCs) are performed annually in the United States and the majority are elective. Current guidelines recommend no fasting prior to elective CC, however recent studies suggest that eating and drinking as desired prior to elective CCs involving moderate sedation is safe.

This project will study the potential benefits of allowing patients to eat before elective CCs. Participants will be randomly divided into two groups. One group will receive pre-op instructions to fast, and the other group will be allowed to eat and drink as desired prior to their CC. Researchers will compare these groups with regards to patient satisfaction and respiratory complications.

ELIGIBILITY:
Inclusion Criteria:

* Willing to comply with all study procedures and remain in contact with the study team to complete study assessments for the duration of the study
* Scheduled for an elective (non-urgent) cardiac catheterization
* Age of 18 or older at the time of consent

Exclusion Criteria:

* Adults unable to consent
* Pregnant women
* Incarceration
* Non-English-speaking patients
* Inability to eat by mouth
* Patients requiring general anesthesia for cardiac catheterization
* Inability to fast for at least 6 hours
* Personal history of pulmonary aspiration, or other known cardiopulmonary anesthetic complication(s)
* Urgent cardiac catheterization
* Inability or unwillingness to comply with all study procedures
* Previously enrolled in this study (patients may not be enrolled more than once for subsequent procedures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2027-09-10 (Estimated); Study Completion 2028-02-10 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | Immediate pre-procedure period, not more than four hours before procedure start-time.
  Six-point ordinal scale response preoperative fasting questionnaire. Self-reported.
Pulmonary aspiration/pneumonitis/pneumonia | From procedure start time to 48 hours post-procedure.
  Indicated by an acute change in oxygen requirement noted in the procedure note or post-procedure progress note. Assessed by chart review. Present/absent.

IPD SHARING:
Plan to Share IPD: Undecided